CLINICAL TRIAL: NCT07346898
Title: Insertion of a Transoesophageal Echocardiography Probe Using McGRATH Video Laryngoscope in Cardiac Surgery Patients: Randomized Controlled Study
Brief Title: Insertion of a Transoesophageal Echocardiography Probe Using McGRATH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Prince Sultan Cardiac Center, Adult Cardiology Department. (Other)
Responsible Party: Principal Investigator, Hassan Mohamed Ali, Professor of anaesthesia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-01-R-096
Record Dates: First submitted 2025-12-19; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Echocardiography, Transesophageal; Cardiac Surgery
Keywords: cardiac anaesthesia, Transesophageal Echocardiography; pharyngeal mucosal injury

STUDY DESIGN:
Intervention Model Description: Prospective, randomized controlled study This is a Parallel-Group Randomized Controlled Trial (RCT) - each participant is randomized into one of two groups, receives only that intervention, and outcomes are compared between groups. There's no crossover, no sequential intervention; both groups proceed in parallel.
  Number of study arms:
  There are two arms:
  Macintosh group (C group) - TEE probe insertion assisted by a conventional Macintosh laryngoscope.
  McGRATH group (M group) - TEE probe insertion assisted by a McGRATH video laryngoscope.
  Each arm receives a distinct intervention, and the primary endpoint (incidence of pharyngeal mucosal injury) will be compared between them.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- McGRATH group (Active Comparator): TEE probe insertion assisted by McGRATH MAC video laryngoscope in an intubated patient under general anesthesia, head in neutral position.
  Interventions: Device: McGRATH group
- Macintoch group (Active Comparator): TEE probe insertion assisted by conventional Macintosh laryngoscope in an intubated patient under general anesthesia, head in neutral position.
  Interventions: Device: Macintosh group

INTERVENTIONS:
Device: McGRATH group — McGRATH video laryngoscope used to assist TEE probe insertion in an intubated patient under general anesthesia
  Other Names: M group
  Arms: McGRATH group
Device: Macintosh group — Macintosh laryngoscope used to assist TEE probe insertion in an intubated patient under general anesthesia
  Other Names: C group
  Arms: Macintoch group

SUMMARY:
This randomized, parallel-group clinical trial compares McGRATH video laryngoscope-assisted versus Macintosh laryngoscope-assisted transoesophageal echocardiography (TEE) probe insertion in adult elective cardiac surgery patients. The primary aim is to compare incidence of pharyngeal mucosal injury during TEE probe insertion.

DETAILED DESCRIPTION:
Transoesophageal echocardiography (TEE) is essential in cardiac anesthesia but TEE probe insertion can cause oropharyngeal mucosal injury and, rarely, esophageal perforation. In this prospective randomized study, adults (≥18 years, ASA II-III) undergoing elective cardiac surgery requiring intraoperative TEE will be randomized 1:1 to TEE probe insertion assisted by either the McGRATH MAC video laryngoscope (M group) or a conventional Macintosh laryngoscope (C group). After induction and tracheal intubation, TEE probe insertion will be attempted with the head in neutral position; the esophageal inlet visibility, number of attempts, total insertion time (seconds), intraoperative vital signs during insertion, and anesthesiologist satisfaction will be recorded. A blinded observer will assess pharyngeal mucosal injury (laceration and/or hematoma) immediately after probe removal. Sample size: 100 (50 per arm). An interim safety analysis will occur after 50 patients; a DSMB will review safety.

ELIGIBILITY:
Inclusion Criteria:

* Adults (male or female) aged ≥ 18 years
* ASA physical status II or III
* Scheduled for elective cardiac surgery under general anesthesia requiring intraoperative transoesophageal echocardiography
* Able to provide written informed consent

Exclusion Criteria:

* Dysphagia or sore throat
* Oropharyngeal infection
* Cervical spine pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of pharyngeal mucosal injury | Immediately after TEE probe removal (intraoperatively)
  Presence of laceration and/or hematoma in the posterior pharyngeal wall, postcricoid area, lateral/medial walls of the piriform sinuses, or the esophageal inlet as observed by a blinded observer after removal of the TEE probe.

SECONDARY OUTCOMES:
Visibility of the oesophageal inlet | During TEE probe insertion (first insertion attempt, intraoperatively)
  Categorical - "Visible" vs "Not visible" as recorded by the operator.
Duration of TEE probe insertion (seconds) | During the intraoperative TEE probe insertion procedure
  Total duration in seconds from mouth opening to successful esophageal insertion, summed across all insertion attempts.
Number of insertion attempts | During the intraoperative TEE probe insertion procedure
  Count of discrete insertions into the mouth until successful esophageal passage or study-defined stop

CONTACTS AND LOCATIONS:
Locations (1):
- Prince Sultan Cardiac Center, Riyadh, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2026-01-07): https://cdn.clinicaltrials.gov/large-docs/98/NCT07346898/Prot_SAP_000.pdf
  • Informed Consent Form (2026-01-07): https://cdn.clinicaltrials.gov/large-docs/98/NCT07346898/ICF_001.pdf